CLINICAL TRIAL: NCT01810094
Title: Prospective Observational Study of Minimally Invasive Fixation of Thoracolumbar Fractures With the Fracture Fixation System S4, Performed With the Fracture Reduction Instrumentation FRI (FRIFIX)
Brief Title: Minimally Invasive Reduction and Fixation of Thoracolumbar Fractures
Acronym: FRIFIX
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-0910
Record Dates: First submitted 2013-02-26; First posted 2013-03-13 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Thoracic Fracture; Lumbar Fracture
Keywords: thoracolumbar fracture; fixation; fixateur interne; minimal invasive; percutaneous
MeSH Terms: conditions — Fractures, Bone | interventions — Fracture Fixation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Minimally invasive Approach: Patients with a thoracolumbar Fracture A3.1 to A 3.3 treated by fracture fixation by a minimally invasive approach
  Interventions: Device: Fracture Fixation

INTERVENTIONS:
Device: Fracture Fixation — Thoracolumbar Fracture Fixation

SUMMARY:
Spinal injuries, such as vertebral fractures, often result in a significant instability of the spine and lead to acute or delayed neurological deficits. Depending on the type of injury there are various methods available to stabilize the spine. The proposed study should clarify whether the combined reduction and fixation with a minimally invasive approach can actually be done with the same precision as in a conventional approach. The primary endpoint of this investigation is the monosegmental anterior wedge angle (AWA), and its maintenance over the first 6 postoperative weeks. It is the aim of the study to gather key radiological, clinical and subjective patient outcome parameters for its patient population that will allow to compare the results to a historical group of patients. The study design is non-interventional, prospective, open,and multicentric.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of the patients of 18 years
* Indication for operative treatment of fractures of the thoracic or lumbar spine
* Singular A3.1-3 fractures according to the AO classification system
* Declaration of consent in participation in this study and willingness to the treatment according to the study protocol
* Physical and mental ability to meet the clinical and radiological follow-up plan

Exclusion Criteria:

* Additional severe trauma, that makes survey of the patient difficult or impossible influence the results of the fracture treatment significantly
* Additional trauma or fractures of the spine
* Other serious conditions complicating participation in the study
* Systemic or local infections
* Pregnancy or planned pregnancy
* Neurological deficits
* Severe blood coagulation disorders diagnosed preoperatively
* Intake of preoperatively anticoagulants
* Osteoporosis
* Bone metabolism disorders
* Laminectomy necessary during surgery results in exclusion of the patient either

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Anterior wedge angle (AWA) | 6 weeks

SECONDARY OUTCOMES:
Blood loss of the patient during surgery to stabilize the spine fracture | intraoperative
OP duration | intraoperative
Adverse events | Intraop and Postop
VAS Spine Score | 3 days and 6 weeks
VAS pain score | 3 days and 6 weeks
accompanying pain medication (or "self medication") | 6 weeks
patient satisfaction with operational results | 6 weeks
  The patient is asked the question whether he is satisfied with the results of the operation, he has the choice between six answers: very satisfied, satisfied, partly satisfied, unsatisfied, no comment
Hospital length of stay | discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hans Goost, MD, Principal Investigator — University Hospital, Bonn
Locations (4):
- Germany (4):
  - Vinzenz-Pallotti-Hospital, Bergisch Gladbach
  - Universitätsklinik Bonn, Abteilung für Unfallchirurgie, Bonn
  - Klinik für Unfall-, Hand- und Wiederherstellungschirurgie, Universitätsklinik Köln, Cologne
  - Abteilung für Orthopädie und Unfallchirurgie, Krankenhaus Wermelskirchen, Wermelskirchen